CLINICAL TRIAL: NCT00325962
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Study of the Effects of 6R-BH4 on Blood Pressure in Subjects With Poorly Controlled Systemic Hypertension
Brief Title: A Study of the Effects of 6R-BH4 on Blood Pressure in Subjects With Poorly Controlled Systemic Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTN-001
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
Keywords: Hypertension; Type 2 Diabetes; 6R-BH4; BH4; BH4 deficiency; sapropterin dihydrochloride; endothelial dysfunction; NO; Nitric Oxide
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Phenylketonurias | interventions — sapropterin

INTERVENTIONS:
Drug: 6R-BH4 (sapropterin dihydrochloride)

SUMMARY:
The purpose of this study is to determine whether 6R-BH4 (sapropterin dihydrochloride) is safe and effective in the treatment of poorly controlled hypertension in the presence or absence of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any research-related procedures.
* At least 18 years of age.
* Willing and able to comply with all study-related procedures.
* History of documented essential hypertension (BP greater than or equal to 140 mm Hg systolic and/or 90 mm Hg diastolic measured on 2 separate occasions).
* Have poorly controlled hypertension despite use of at least two conventional antihypertensive agents with different mechanisms of action taken concurrently and consistently for at least 3 months before randomization. (Note: Antihypertensive agents may be individual or combined into a single medication.)
* During the two-week screening period, mean SBP and mean DBP fall within the following ranges:
* Mean SBP between 135 and 160 mm Hg
* Mean DBP between 85 and 110 mm Hg
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
* Females of childbearing potential must have a negative pregnancy test at screening and be willing to have additional pregnancy tests during this study.

Individuals in the diabetic cohort must meet this additional criterion:

* Documented history of type 2 diabetes that has been treated using the same therapy for at least 3 months.

Exclusion Criteria:

* Previous treatment with any formulation of BH4.
* Known allergy or hypersensitivity to any excipient of 6R-BH4.
* Known secondary cause for hypertension.
* Concurrent disease or condition that would interfere with study participation or safety such as bleeding disorders, history of syncope or vertigo, severe gastrointestinal reflux disease (GERD), symptomatic coronary or peripheral vascular disease, arrhythmia, organ transplant, organ failure, or type 1 diabetes mellitus.
* Any sever co-morbid condition that would limit life expectancy to less than 6 months.
* Serum creatinine >2.0mg/dL or hepatic enzyme levels more than 2 times the upper limit of normal.
* Requirement for concomitant treatment with any drug known to inhibit folate metabolism (e.g., methotrexate).
* Concomitant treatment with levodopa.
* Concomitant treatment with any phosphodiesterase (PDE) 5 inhibitor (e.g., Viagra(R), Cialis(R), or Levitra(R), or Revatio (TM) or any PDE 3 inhibitor (e.g., cilostazol, milrinone, or vesnarinone).)
* Use of any investigational product or device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Pregnant or breastfeeding at screening or planning to become pregnant (subject or partner) at any time during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2006-05; Primary Completion 2006-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To compare oral 6R-BH4 to placebo with respect to change from baseline in arterial systolic blood pressure after 8 weeks of treatment in subjects with poorly controlled hypertension.

SECONDARY OUTCOMES:
To compare oral 6R-BH4 to placebo with respect to change from baseline in arterial diastolic blood pressure after 8 weeks of treatment in subjects with poorly controlled hypertension
To compare oral 6R-BH4 to placebo with respect to change from baseline in insulin sensitivity after 8 weeks of treatment in subjects with both type 2 diabetes and poorly controlled hypertension
To compare oral 6R-BH4 to placebo with respect to change from baseline in eNOS activity and endothelial dysfunction after 8 weeks of treatment in subjects with poorly controlled hypertension
To assess the safety of oral dosing of 6R-BH4 in subjects with poorly controlled hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Martha Nicholson, MD, Study Director — BioMarin Pharmaceutical
Locations (24):
- United States (24):
  - Hoover, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Muscle Shoals, Alabama
  - Gilbert, Arizona
  - Phoenix, Arizona
  - Anaheim, California
  - Burbank, California
  - Cudahy, California
  - Long Beach, California
  - Roseville, California
  - San Francisco, California
  - Denver, Colorado
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Indianapolis, Indiana
  - Auburn, Maine
  - Scarborough, Maine
  - Baltimore, Maryland
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Knoxville, Tennessee
  - Carrollton, Texas

REFERENCES:
- See also: BioMarin Pharmaceutical Inc. website — http://www.bmrn.com